CLINICAL TRIAL: NCT03215615
Title: Evaluation of Two Resin Composites and Two Adhesives for a Novel Surgical-restorative Protocol for the Treatment of Non-carious Cervical Lesions Associated With Gingival Recession: a Randomized Controlled Clinical Trial
Brief Title: Evaluation of Two Resin Composites and Two Adhesives for a Novel Restorative Protocol to Treat Cervical Lesions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Responsible Party: Principal Investigator, Eduardo Bresciani, Associate Professor, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 56450116.9.0000.0077
Record Dates: First submitted 2016-11-24; First posted 2017-07-12 (Actual); Last update posted 2019-06-13 (Actual); Status verified 2019-06

CONDITIONS: Dental Abrasion; Gingival Recession; Composite Resins
MeSH Terms: conditions — Tooth Abrasion; Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group NF + TE (Active Comparator): Nanofilled Composite - Filtek Z350 XT® - 3M ESPE (NF) + Total Etch adhesive - Adper Single Bond 2® - 3M ESPE (TE) adhesive: combined lesions will be treated with partial restoration with nanofilled resin composite and total-etch adhesive system (two step). Subsequently, periodontal surgery will be performed for root coverage.
  Interventions: Procedure: Periodontal surgery; Procedure: Total Etch adhesive; Procedure: Nanofilled Composite
- Group NF + UA (Active Comparator): Nanofilled Composite - Filtek Z350 XT® - 3M ESPE (NF) + Universal Adhesive - Single Bond Universal® - 3M ESPE (UA): combined lesions will be treated with partial restoration with nanofilled resin composite and one-step self-etching adhesive system. Subsequently, periodontal surgery will be performed for root coverage.
  Interventions: Procedure: Periodontal surgery; Procedure: Universal Adhesive; Procedure: Nanofilled Composite
- Group MH + TE (Active Comparator): Micro-Hybrid Composite - Charisma Classic® - Heraeus Kulzer (MH) + Total Etch adhesive - Adper Single Bond 2® - 3M ESPE (TE) adhesive: combined lesions will be treated with partial restoration with micro-hybrid resin composite and total-etch adhesive system (two step). Subsequently, periodontal surgery will be performed for root coverage.
  Interventions: Procedure: Periodontal surgery; Procedure: Total Etch adhesive; Procedure: Micro-Hybrid Composite
- Group MH + UA (Active Comparator): Micro-Hybrid Composite - Charisma Classic® - Heraeus Kulzer (MH) + Universal Adhesive - Single Bond Universal® - 3M ESPE (UA): combined lesions will be treated with partial restoration with micro-hybrid resin composite and one-step self-etching adhesive system. Subsequently, periodontal surgery will be performed for root coverage.
  Interventions: Procedure: Periodontal surgery; Procedure: Universal Adhesive; Procedure: Micro-Hybrid Composite

INTERVENTIONS:
Procedure: Periodontal surgery — Coronally advanced flap for root coverage
Procedure: Total Etch adhesive — Total-etch adhesive system (two step)
  Arms: Group MH + TE; Group NF + TE
Procedure: Universal Adhesive — One-step self-etching adhesive system
  Arms: Group MH + UA; Group NF + UA
Procedure: Nanofilled Composite — Partial nanofilled-resin composite restoration
  Arms: Group NF + TE; Group NF + UA
Procedure: Micro-Hybrid Composite — Partial micro-hybrid composite restoration
  Arms: Group MH + TE; Group MH + UA

SUMMARY:
Non-carious cervical lesion is frequently associated with gingival recession, resulting in a combined lesion that has a different treatment prognosis when the two lesions appear alone. The literature presents few studies that propose a multidisciplinary approach (restorative and root coverage surgery procedures) to optimize the treatment of this combined lesion. The previously proposed approaches and materials have limitations and an optimal clinical protocol has not been established yet. Thus the aim of this study is to evaluate a novel multidisciplinary protocol with two resin composites and two different adhesive systems through a randomized clinical trial and laboratory studies. 120 combined lesions will be randomly assigned to one of the following groups: NP + TE (n = 30) - Partial restoration of cervical lesions with nanofilled composite and total-etch adhesive system and periodontal surgery for root coverage, NP + UA (n = 30) - partial restoration of cervical lesions with nanofilled composite and self-etching adhesive system and periodontal surgery for root coverage, MH + TE (n = 30) - partial restoration of cervical lesions with microhybrid composite and total-etch adhesive system and periodontal surgery for root coverage, MH + UA (n = 30) - partial restoration of cervical lesions with microhybrid composite and self-etching adhesive system and periodontal surgery for root coverage. Restorations will be assessed using the USPHS criteria after one week, six months and twelve months.

ELIGIBILITY:
Inclusion Criteria:

* Individuals presenting one or more combined defect, i.e. a NCCL classified as B+ (Pini-Prato et al., 2010): presenting more than 1mm in depth, affecting dental crown and root associated with Miller's class I or II gingival recession in canines or premolars with pulp vitality;
* Healthy patients (systemically and periodontally), 18 years old, with at least 20 teeth in occlusion;
* Plaque index ≤ 20% (Ainamo & Bay, 1975);
* NCCL cavo-surface margin without involvement of more than 50% of enamel;
* In tooth included in the study and the adjacent elements of the following must be observed: probing depth less than 3 mm; do not show bleeding on probing (periodontal health) and no insertion loss in the proximal and palatal areas; Provide formal consent to participate in research, after the explanation of the risks and benefits by an individual not involved in it (Resolution #196 October 1996 and the Code of Dental Professional Ethics - C.F.O. - 179/93).

Exclusion Criteria:

* NCCL previously restored;
* Presence of caries;
* Patients with periodontitis;
* Patients with bruxism or teeth clenching;
* Patients with orthodontic treatment in progress;
* Pregnant patients or smokers;
* Patients with systemic problems (cardiovascular, blood dyscrasias, immunodeficiency, diabetes and others), which contraindicate the surgical procedure; Previous periodontal surgery in the area of interest of the present study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-11; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Modified United States Public Health Service (USPHS) criteria | 1 year
  USPHS criteria is based on the following ratings: Color compatibility, retention, marginal adaptation, anatomic form, surface texture, marginal discoloration, sensibility pre-operative and postoperative and the presence of secondary caries

SECONDARY OUTCOMES:
Aesthetics (Visual Analogue Acale - VAS) | 1 year
  The esthetics of the treatment will be evaluated by patients´ point of view using the VAS scale
Dentin Hypersensitivity (Visual Analogue Acale - VAS) | 1 year
  The Dentin Hypersensitivity will be evaluated by patients´ point of view using the VAS scale

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Bresciani, PhD, Principal Investigator — Universidade Estadual Paulista Júlio de Mesquita Filho
Locations (1):
- UEPJMF, São José dos Campos, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mathias-Santamaria IF, Santamaria MP, Silveira CA, Martinho FC, de Melo MAS, De Marco AC, Augusto MG, de Andrade GS, Roulet JF, Bresciani E. Evaluation of a novel restorative protocol to treat non-carious cervical lesion associated with gingival recession: a 2-year follow-up randomized clinical trial. Clin Oral Investig. 2023 Apr;27(4):1781-1792. doi: 10.1007/s00784-022-04806-1. Epub 2022 Dec 3. PMID 36462038